CLINICAL TRIAL: NCT05472649
Title: Long-Term Follow-Up Study of Patients Who Have Received Gene-Modified Cell Therapy or Gene Therapy in Trials Sponsored By Sorrento Therapeutics, INC.
Brief Title: Long-Term Follow-Up of Patients Who Received Gene-Modified Cell Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CGT-LTFU-351
Record Dates: First submitted 2022-07-13; First posted 2022-07-25 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Long-term Follow-up
Keywords: long-term follow up

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants exposed to Gene-Modified Cell Therapy
  Interventions: Biological: Gene-Modified Cell Therapy

INTERVENTIONS:
Biological: Gene-Modified Cell Therapy — No investigational cell product will be administered

SUMMARY:
Observational long-term follow-up study of patients who have been exposed to a gene-modified cell therapy produced by ex vivo transduction of immune cells expressing viral or non-viral vectors in studies sponsored by Sorrento Therapeutics, Inc.

DETAILED DESCRIPTION:
Study CGT-LTFU-35 is an observational study of patients who have been exposed to a gene-modified cell therapy (GMCT) produced by ex vivo transduction of immune cells expressing viral and/or non-viral vectors in studies sponsored by Sorrento Therapeutics, Inc. Patients are to be followed for up to 15 years after exposure to a GMCT agent for the possible development of long-term adverse events and efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received any amount of a CGT in a study sponsored by Sorrento Therapeutics, Inc.

Exclusion Criteria:

* Unable or unwilling to provide written informed consent and/or comply with study requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were exposed to gene-modified cell therapy produced by ex vivo transduction of immune cells expressing viral or non-viral vectors in studies sponsored by Sorrento Therapeutics, Inc.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2036-12 (Estimated); Study Completion 2037-05 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of previous treatment with gene-modified cells | Baseline through end of study (approximately 15 years)
  Long-term safety of previous treatment as assessed by incidence of adverse events (AEs)

SECONDARY OUTCOMES:
Long-term durability of clinical effect of previous treatment with gene-modified cells | Baseline through end of study (approximately 15 years)
  Long-term durability of clinical effect of previous treatment with gene-modified cells as assessed by duration of response (DOR)
Long-term durability of previous treatment with gene modified cells | Baseline through end of study (approximately 15 years)
  Long-term durability as assessed by progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (1):
- Abramson Cancer Center Clinical Research Unit, University of Pennsylvania, Philadelphia, Pennsylvania, United States